CLINICAL TRIAL: NCT06144866
Title: Evaluation of Non-Vitamin K Antagonist Oral Anticoagulants Concentration Among Patients With Acute Stroke (The Direct Oral AntiCoagulant Registry in Taiwan-Emergent Department, DOACT-ED)
Brief Title: Evaluataion of NOAC Levels in Acute Stroke
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Principal Investigator, National Taiwan University Clinical Trial Center, Pharmacist, National Taiwan University Hospital
Other Study IDs: 202003059RINA
Record Dates: First submitted 2023-11-17; First posted 2023-11-22 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Ischemic Stroke; Anticoagulant Adverse Reaction
Keywords: Ischemic stroke; Intracranial hemorrhage; Direct oral anticoagulant; Drug level
MeSH Terms: conditions — Ischemic Stroke; Intracranial Hemorrhages | interventions — Dabigatran; Rivaroxaban; apixaban; edoxaban; N(4)-oleylcytosine arabinoside

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — plasma, buffycoat
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Dabigatran, rivaroxaban, apixaban, edoxaban — For patients who received direct oral anticoagulants (DOAC) before ischemic stroke or intracranial hemorrhage, the DOAC level upon hospital arrival will be measured.
  Other Names: Direct oral anticoagulants

SUMMARY:
Non-vitamin K antagonist oral anticoagulants (NOACs) are recommended over warfarin in preventing stroke and thromboembolism among patients with atrial fibrillation (AF) in several guidelines. To evaluate the pharmacological effects of NOACs, directly measuring the concentration is the most arbitrary way since the correlation between concentration and common coagulation tests are not reliable. Our previous investigation reported under the fixed dose regimen, dabigatran exposure increased in elderly, renal impairments and patients with multiple co-morbid conditions. Our data also showed difference in NOACs exposure in Asians. For example, patients under rivaroxaban, in comparison to apxiaban, were more likely to have lower than expected range drug level. Furthermore, the NOACs concentration also affected by the prescription pattern of physicians (non-compliant to labeled dose) and patients' behavior (poor medication adherence).

The relationship between NOACs exposure and safety has been elucidated in large-scale clinical trials. As the NOACs level increased, the risk for bleeding increased, too. Nevertheless, no additional protection was noted with increased NOACs levels. In post marketing surveillance, bleeding and thrombotic events have been reported. Investigating the NOACs level among these patients helps evaluating the residual drug in the body, which could be a reference for clinical decision in emergent situation.

Specific purpose: Investigate the correlation between NOACs concentration upon the arrival of emergency department (ED) and important clinical outcomes including systemic thromboembolism, and major bleeding.

Direction for investigation:

1. Prospectively record the NOACs concentration among AF patients under NOACs therapy and suffered from ischemic stroke (IS), transient ischemic attack (TIA), intracerebral hemorrhage (ICH) and other major bleeding.
2. Investigate the correlation between NOACs concentration upon ED arrival and thromboembolic or bleeding events.
3. Propose a therapeutic range for NOACs, in order to provide a guide for important decision in acute setting.

DETAILED DESCRIPTION:
Non-vitamin K antagonist oral anticoagulants (NOACs) are recommended over warfarin in preventing stroke and thromboembolism among patients with atrial fibrillation (AF) in several guidelines. To evaluate the pharmacological effects of NOACs, directly measuring the concentration is the most arbitrary way since the correlation between concentration and common coagulation tests are not reliable. Our previous investigation reported under the fixed dose regimen, dabigatran exposure increased in elderly, renal impairments and patients with multiple co-morbid conditions. Our data also showed difference in NOACs exposure in Asians. For example, patients under rivaroxaban, in comparison to apxiaban, were more likely to have lower than expected range drug level. Furthermore, the NOACs concentration also affected by the prescription pattern of physicians (non-compliant to labeled dose) and patients' behavior (poor medication adherence).

The relationship between NOACs exposure and safety has been elucidated in large-scale clinical trials. As the NOACs level increased, the risk for bleeding increased, too. Nevertheless, no additional protection was noted with increased NOACs levels. In post marketing surveillance, bleeding and thrombotic events have been reported. Investigating the NOACs level among these patients helps evaluating the residual drug in the body, which could be a reference for clinical decision in emergent situation.

Specific purpose:

1. Prospectively record the NOACs concentration among AF patients under NOACs therapy and suffered from IS, TIA, ICH or major bleeding.

   AF patients who presented to emergent department (ED) for acute IS, TIA, ICH (non-traumatic), or other major bleeding and was under NOACs therapy will be recruited to this study. Blood sample will be collected before acute management to measure NOACs concentration. Co-morbid disease, laboratory tests and concurrent medications will be retrieved from electronic medical records. The onset, location, severity of IS. ICH or other major bleeding, and the outcome and long-term managements will be prospectively recorded.
2. Investigate the correlation between NOACs concentration and thromboembolic or bleeding events.

   For each NOACs, we are going to compare the differences in NOACs exposure between patients with thromboembolism or major bleedi. Important baseline characteristics, co-medications and disease severity will be adjusted before making comparison.
3. Propose a therapeutic range for NOACs, in order to provide a guide for important decision in acute setting.

From the data of NOACs concentration among patients with IS or ICH, we plan to propose a therapeutic range with acceptable efficacy and safety for NOACs therapy. Our data will provide a guide for physicians to make important clinical decision.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 20 years
2. Having AF diagnosis
3. Under NOACs therapy including dabigatran, rivaroxaban, apixaban and edoxaban.
4. Admitted for acute IS, transient ischemic attack (TIA), ICH or major bleeding

Exclusion Criteria:

1. The ICH is resulted from trauma.
2. Decline the inform consent.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient under direct oral anticoagulant therapy and suffered from ischemic stroke or intracranial hemorrhage.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Functional outcome | 3 months after stroke (ischemic or hemorrhagic)
  Functional status measured by using the modified Rankin Scale.

SECONDARY OUTCOMES:
Symptomatic intracranial hemorrhage (sICH) | 24-36 hours after stroke
  Type 2 parenchymal hemorrhage on the follow-up neuroimage in 24 to 36 hours after EVT, with neurological deterioration of ≥4 points on the National Institute of Health Stroke Scale (NIHSS) score from baseline
Early neurological improvement | 24 hours after stroke
  Reduction of 8 points or more in the NIHSS score within 24 hours.
Successful reperfusion (in ischemic stroke patients receiving endovascular thrombectomy) | Evaluated after EVT
  Defined as Thrombolysis in Cerebral Infarction (TICI) scale 2b to 3
Recurrent ischemic stroke | 3 years
  Neurological symptoms with ischemic lesion noted on neuroimaging
Recurrent intracranial hemorrhage | 3 years
  Neurological symptoms with hemorrhagic lesion noted on neuroimaging

CONTACTS AND LOCATIONS:
Overall Officials: Shin Yi Lin, M.S., Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No